CLINICAL TRIAL: NCT01208987
Title: Improving Laboratory Follow-up by Delivering an Enhanced Medication List to Outpatient Physician Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0710-59
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Medication Histories in Outpatient Clinic Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (with Medication History) (Experimental): these patient visits generated a medication history
  Interventions: Other: Medication History was printed

INTERVENTIONS:
Other: Medication History was printed

SUMMARY:
The investigators plan to develop a process to create an Enhanced Medication List. The INPC (Indiana Network for Patient Care) already obtains histories of medications dispensed by pharmacies from several sources: pharmacy benefit managers, RxHub, insurance companies, Medicaid, SureScripts, Wishard Health Services. The investigators will collect all the medication data available through the INPC for an individual patient. The investigators will enhance this medication list by including medication categories, improving the structure and appearance, displaying results of relevant laboratory tests, and adding decision support reminders. The investigators will test the value of such an "Enhanced Medication List" by providing it to outpatient physician practices (through the DOCS4DOCS clinical messaging service, or as a fax), preferably on the day that the patient has an office visit with the physician. The investigators will determine whether this intervention improves patient care: whether there are higher rates of recommended laboratory follow-up monitoring as a result; whether there are lower rates of harmful drug-drug interactions. The investigators will also seek the opinions of physicians regarding the benefit of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* outpatient clinic patient visits

Exclusion Criteria:

* Age 18 and under

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5256 (Actual)
Dates: Start 2007-09-28 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-01 (Actual)

PRIMARY OUTCOMES:
Count of medications (on a patient's medication list) for which recent (within 12 months) laboratory test monitoring is missing. | Laboratory tests during the previous 12 months
  The hypothesis is that the intervention (a medication history printed for the patient) would help the physician identify incomplete monitoring of laboratory test results for a subset of medications. (For example, Potassium test levels should be obtained every 12 months for patients using diuretics, according to NCQA HEDIS guidelines.) With time, the intervention group should have less medications for which laboratory test results are incomplete. Therefore, the intervention group should have less medications with decision support reminders warning of incomplete laboratory test monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenstrief Institute, Indianapolis, Indiana, United States